CLINICAL TRIAL: NCT05906576
Title: Post-marketing Registry Study of Infliximab for Injection in Chinese Pediatric Crohn's Disease Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Taizhou Mabtech Pharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C008CDIV
Record Dates: First submitted 2023-06-02; First posted 2023-06-18 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Infliximab (Experimental): Infliximab for the treatment of Crohn's disease in children
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab — Infliximab in the treatment of Crohn's disease in children
  Other Names: CMAB008

SUMMARY:
Post-marketing registration of Infliximab for injection in Chinese pediatric Crohn's disease patients.

DETAILED DESCRIPTION:
This is a prospective, multicenter registry study in Chinese pediatric Crohn's disease patients. A total of 30 subjects were planned to be enrolled and treated with Infliximab. Subjects were observed for 102 weeks after administration to evaluate the clinical efficacy and safety of infliximab in the treatment of children with Crohn's disease in a real diagnostic setting.

ELIGIBILITY:
Inclusion Criteria:

1. Age ranged 6 to 17 years (both inclusive), no gender limitation.
2. A clear diagnosis was made in children with moderate to severe active stage (PCDAI≥30) Crohn's disease refer to the expert consensus on the diagnosis and treatment of inflammatory bowel disease in children (2019 edition).
3. Patients and/or their guardians must sign ICF, and the research agreement/ICF for data collection and data verification shall comply with local laws and regulations.
4. The patient received infliximab for the first time.

Exclusion Criteria:

1. Patients with contraindications to infliximab use (such as severe infection, active tuberculosis, lymphoma or other malignancies), moderate to severe heart failure, and allergies to other murine proteins, infliximab or any component of this product.
2. Those who accept other anti-TNF-α any biological drugs or any other biologicals.
3. Patients who plan to receive live vaccine within 3 months before signing the informed consent or during the treatment period
4. Those who have been or being enrolled in other clinical studies within 3 months prior to signing ICF
5. The investigator judges the subject inappropriate to be included in this study.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Clinical response rate at 14 weeks | up to 14 weeks
  Clinical response: PCDAI decreased ≥15 points and total PCDAI≤ 30 points

SECONDARY OUTCOMES:
Clinical remission rate at week 14 and 54 | up to 54 weeks
  Clinical remission: PCDAI≤10
Endoscopic response rate at week 14 and 54 | up to 54 weeks
  Endoscopic response: SES-CD decreased ≥ 50%
Mucosal healing rate at week 14 and 54 | up to 54 weeks
  Mucosal healing: SES-CD 0-2
Changes from baseline in height-for-age z-score (HAZ), weight-for-age z-score (WAZ) and BMI-for-age z-score at week 14 and 54 | up to 54 weeks
  The z-score is converted from anthropometric measurements based on the World Health Organization growth reference. The z-score including: height-for-age z-score (HAZ), weight-for-age z-score (WAZ) and BMI-for-age z-score.
Changes from baseline in serum C-reactive protein at week 14 and 54 | up to 54 weeks
  Changes from baseline in serum C-reactive protein at week 14 and 54
Changes from baseline in erythrocyte sedimentation rate at week 14 and 54 | up to 54 weeks
  Changes from baseline in erythrocyte sedimentation rate at week 14 and 54
Changes from baseline in the rate of delayed development of adolescents at 14 and 54 weeks | up to 54 weeks
  Delayed development: Female children over 13 years old and male children over 14 years old are in the Tanner stage I
ADA positive rate | up to 54 weeks
  ADA positive rate at week 14 and 54
Percentage of participants with Adverse Events | up to 102 weeks
  Total Frequency of Adverse Events/Serious Adverse Events Within the Whole Time of the Study

CONTACTS AND LOCATIONS:
Overall Officials: Wu Jie, Principal Investigator — Beijing Children's Hospital
Locations (1):
- Beijing Children's Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No